CLINICAL TRIAL: NCT06429982
Title: A Clinical Trial to Assess Whether Dexamethasone Addition to Standard Protocols for Non-Traumatic Rhabdomyolysis of Unknown or Genetic Etiologies Improves Patient Outcomes
Brief Title: Dexamethasone Use in Pediatric Rhabdomyolysis Patients in Addition to Standard Protocols
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Natasha Shur, MD, Principal Investigator, Professor, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000710
Record Dates: First submitted 2023-08-31; First posted 2024-05-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis | interventions — Dexamethasone; Sugars

STUDY DESIGN:
Intervention Model Description: There will be a 2: 1 treatment ratio of dexamethasone treated group versus placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be double-blinded. The pharmacy will determine which patients are in the study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone group (Active Comparator): Dexamethasone five days with 0.6 mg/ kg dose per day max 16 mg dose. Standard care will also be provided.
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): Placebo for five days with one dose per day placebo oral dosing. Standard care will also be provided.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Steroid five day treatment
  Other Names: DexPak
  Arms: Dexamethasone group
Drug: Placebo — Placebo control group
  Other Names: Sugar Pill
  Arms: Placebo group

SUMMARY:
There is a significant unmet need for optimized treatment in rhabdomyolysis. There are few prospective interventional studies on treatment for rhabdomyolysis, a condition which affects diverse and underrepresented populations at a higher rate. While steroids are often used off-label, a systematic study has not yet been initiated, and steroids have not been yet considered in as a consideration to standard care guidelines.

The hypothesis is that patients who receive dexamethasone in addition to standard care versus placebo and standard care will have improvement in pain, length of hospital stay, and decrease in kidney complications.

DETAILED DESCRIPTION:
Study Objective:

This is a single center, 2-year, blinded prospective randomized study for those diagnosed with rhabdomyolysis age six months-25 years using dexamethasone versus placebo treatment in addition to standard care in up to 50 patients.

Study Design:

Patients will be enrolled with a 2:1 ratio of treatment of dexamethasone for 5 days versus placebo treatment for 5 days in addition to receiving standard care. The treatment period for each subject will be five days treatment with oral treatment once per day with study drug (dexamethasone versus placebo). All patients will also receive standard care. Patients and their parent/ caregiver will have the option to complete surveys before and after treatment in order to assess pain level and treatment improvement. Chart review will be performed on all patients throughout and after the five-day study treatment period. There will be no additional interventions.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of rhabdomyolysis defined as creatine kinase> 5000 with trauma excluded
2. Ability of parents/patients to understand and the willingness to sign a written informed consent document.
3. Patients ages 12 and older will sign written assent

Exclusion Criteria:

* Already taking systemic steroids.
* Inability to comply with study instructions.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women.

  o A urine pregnancy test will be performed for women of child-bearing potential.
* Below gestational age of 40 weeks
* Allergy to fluconazole, clotrimazole or nystatin.
* Cannot tolerate PO medications

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | Primarily 5 days - 1 year
  Number of days Length of Stay in Each Group
Muscle breakdown | Primarily 5 days - 1 year
  Creatinine Kinase trend comparison between groups
Renal complications | Primarily 5 days - 1 year
  Bun/ Creatinine

SECONDARY OUTCOMES:
Quantitative Pain Outcomes | 14 days
  EHR pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Shur, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chavez LO, Leon M, Einav S, Varon J. Beyond muscle destruction: a systematic review of rhabdomyolysis for clinical practice. Crit Care. 2016 Jun 15;20(1):135. doi: 10.1186/s13054-016-1314-5. PMID 27301374
- [Background] Summerlin ML, Regier DS, Fraser JL, Chapman KA, Kafashzadeh D, Billington C Jr, Kisling M, Grochowsky A, Ah Mew N, Shur N. Use of dexamethasone in idiopathic, acute pediatric rhabdomyolysis. Am J Med Genet A. 2021 Feb;185(2):500-507. doi: 10.1002/ajmg.a.62000. Epub 2020 Dec 10. PMID 33300687
- [Background] Szugye HS. Pediatric Rhabdomyolysis. Pediatr Rev. 2020 Jun;41(6):265-275. doi: 10.1542/pir.2018-0300. PMID 32482689